CLINICAL TRIAL: NCT03255122
Title: Harnessing Technology to Extend the Reach of Supported Care for Families Affected by Early Child Social Anxiety
Brief Title: Technology and Early Anxiety Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Andrew Kukes Foundation for Social Anxiety (Unknown)
Responsible Party: Principal Investigator, Jonathan S. Comer, Professor of Psychology, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-16-0182
Record Dates: First submitted 2017-03-20; First posted 2017-08-21 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Families are randomly designed to receive either immediate treatment (I-CALM) or waitlist and then I-CALM
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators masked to each participating family's treatment condition will perform all structured diagnostic interviews and generate responder status data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): Individuals in this condition will immediately receive I-CALM treatment, which draws on videoconferencing to remotely deliver real time cognitive-behavioral therapy for early child anxiety to families in their home.
  Interventions: Behavioral: I-CALM
- Waitlist (Other): Individuals in Waitlist will participate in an initial waitlist condition, and then after post-waitlist assessment will be offered the I-CALM intervention. Accordingly families in this condition receive Delayed I-CALM.
  Interventions: Behavioral: Delayed I-CALM

INTERVENTIONS:
Behavioral: I-CALM — Families receiving I-CALM will immediately receive a videoconferencing-based, Internet-delivered format of an evidence-based CBT treatment for early child social anxiety disorder (Coaching Approach behavior and Leading by Modeling, or the CALM Program; Puliafico, Comer, & Albano, 2013) in which therapists and families meet in real-time via videoconferencing and parent-child interactions are broadcast from the family's home via a webcam while therapists provide bug-in-the-ear coaching from a remote site. Parents are taught and guided in how to coach their young anxious child to engage in brave, approach behavior.
  Arms: Immediate treatment
Behavioral: Delayed I-CALM — Families receiving Delayed I-CALM will participate in a waitlist period, and then will complete the I-CALM treatment program.
  Arms: Waitlist

SUMMARY:
The goal of the study is to evaluate the efficacy of an Internet-delivered format of an evidence-based CBT treatment for early social anxiety disorder (Coaching Approach behavior and Leading by Modeling, or the CALM Program) in which therapists and families meet in real-time via videoconferencing and parent-child interactions are broadcast from the family's home via a webcam while therapists provide bug-in-the-ear coaching from a remote site. In a randomized controlled trial (RCT), the proposed work will evaluate 40 youth with social anxiety disorder (ages 3-8); 20 will receive the CALM Program over the Internet (I-CALM) and 20 will be assigned to a waitlist control and will complete a course of I-CALM after the waitlist period. Outcomes will be assessed via structured diagnostic interviews and parent-report questionnaires.

DETAILED DESCRIPTION:
The goal of the study is to evaluate the efficacy of an Internet-delivered format of an evidence-based CBT treatment for early child social anxiety disorder (Coaching Approach behavior and Leading by Modeling, or the CALM Program) in which therapists and families meet in real-time via videoconferencing and parent-child interactions are broadcast from the family's home via a webcam while therapists provide bug-in-the-ear coaching from a remote site. In a randomized controlled trial (RCT), the proposed work will evaluate 40 youth with social anxiety disorder (ages 3-8); 20 will receive the CALM Program over the Internet (I-CALM) and 20 will be assigned to a waitlist control, followed by I-CALM treatment.

SPECIFIC AIMS:

* Aim 1: To evaluate I-CALM efficacy for reducing early child social anxiety symptoms and related impairments and for improving child and parent quality of life.
* Aim 2: To examine the extent to which I-CALM helps families overcome traditional barriers to effective care, including geographic barriers and regional professional workforce shortages in social anxiety expert care.
* Aim 3: To evaluate the feasibility, acceptability, and satisfaction of I-CALM from the perspective of treated\ families, and lay the foundation for a large Florida statewide implementation of I-CALM for early social anxiety.

RATIONALE: Despite progress in supported programs for child social anxiety disorder, gaps persist between treatment in specialty clinics and services broadly available in the community. Although considerable advances show social anxiety is treatable when appropriate CBT is available, barriers interfere with the broad provision of quality care. Few sufferers receive services, and those who do receive services do not necessarily receive evidence-based care. Many U.S. counties have no psychologist, psychiatrist, or social worker, let alone professionals trained in supported social anxiety treatments. When effective programs are available, transportation issues constrain access, with large proportions of patients reporting that services are too far away or they have no way to get to a clinic. Expert providers cluster around metropolitan regions and major academic hubs, leaving considerable numbers of youth without access to supported service options. Youth from low-income or remote and rural communities are particularly unlikely to receive appropriate care. High rates of stigma-related beliefs further constrain service utilization, with many reporting negative attitudes about visiting a mental health clinic.

An Internet-delivered, real-time intervention for the remote treatment of early child social anxiety disorder has the potential to meaningfully extend the reach of effective social anxiety treatment for underserved youth and can serve as the critical foundation upon which to build a larger-scale statewide implementation of early social anxiety treatment. Moreover, treating youth in their homes can overcome stigma-related concerns that interfere with families attending services at a psychiatric clinic, and treatment gains may be more generalizable and ecologically valid as services are provided to youth in their natural settings.

SERVICES: The CALM Program (Coaching Approach behavior and Leading by Modeling) was developed as a developmentally compatible intervention to treat anxiety disorders in children below age 8. The CALM Program is an adaptation of Parent-Child Interaction Therapy (PCIT), which was initially developed to treat early behavior problems, and incorporates a family-based approach to early child anxiety. Whereas effective treatment for older socially anxious youth requires a set of cognitive abilities that younger children typically do not fully possess, it has been demonstrated that adaptations of PCIT-which do not target children directly, but rather work to reshape the primary contexts of child development in order to treat child anxiety-can offer more developmentally compatible approaches for intervening with early social anxiety. The CALM Program is a parent-focused treatment that educates families about social anxiety and teaches parents skills to effectively reinforce their children's brave social behavior and coaches the use of these skills during in-session parent-child interactions. The treatment emphasizes live, bug-in-the-ear coaching of parents during in vivo exposure sessions. Child symptoms are targeted by reshaping interaction patterns associated with the maintenance of child anxiety and by reducing parental accommodation of child bids to avoid social situations.

Traditionally, the CALM therapist is situated behind a one-way mirror and unobtrusively provides real-time feedback to parents through a parent-worn earpiece. It has been suggested that PCIT-based approaches are particularly amenable to a web format given that by design the therapist conducts live observation and feedback from another room via a parent-worn bug-in-the-ear device. That is, even in standard clinic-based CALM, the therapist is predominantly separated from the family in order to foster naturalistic family interactions and child behavior. Despite progress in the development of the CALM Program for social anxiety, and progress in the field of behavioral telehealth, research has yet to evaluate the efficacy of an Internet-delivered format of the CALM Program (I-PCIT) for extending the accessibility of treatment. I-CALM families will receive treatment using secure and encrypted videoconferencing software, and parents will receive live coaching via a Bluetooth earpiece. Independent evaluators will conduct diagnostic interviews, collect parent-report forms, and conduct structured observations at baseline, post-treatment, and 6-months follow-up.

OUTCOMES: Independent evaluators (IEs) masked to participant condition assignment will conduct diagnostic interviews, collect parent-report forms, and conduct structured observations at baseline, post-treatment, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-8 years old, and at least one primary caregiver
* Child has diagnosis of social anxiety disorder (as assessed in pre-treatment assessment).
* Child and parent both speak either English or Spanish fluently
* Family's home is equipped with computing device and high-speed internet

Exclusion Criteria:

* Child has emotional/behavioral problem more impairing than difficulties captured by an anxiety disorder diagnosis.
* Child receiving medication or other psychotherapy to manage emotional difficulties
* History of severe physical or mental impairments (e.g., intellectual disability, deafness, blindness, pervasive developmental disorder) in child or participating caregiver(s)
* Child is a ward of the state

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions Scales - Severity and Improvement (CGI-S/I) | 5 minutes
  CGI-S/I is the most widely used clinician-rated measure of treatment-related changes in functioning (Guy & Bonato, 1970) and will be completed by IEs in the present study. The CGI-S score rates illness severity on a 7-point scale, ranging from 1 ("normal") to 7 ("among the most severely ill patients"). The CGI-I rates clinical improvement on a 7-point scale, ranging from 1 ("very much improved") to 7 ("very much worse").

SECONDARY OUTCOMES:
Children's Global Assessment Scale | 5 minutes
  The Children's Global Assessment Scale (CGAS; Shaffer et al., 1983) is a widely used measure of overall child disturbance, providing a clinician-rated index of functioning. Scores range from 0-100, with lower scores indicating greater functional impairments.
Child Anxiety Impact Scale | 5 minutes
  The Child Anxiety Impact Scale (CAIS) is a brief parent-report measure of anxiety-related functional impairment, and has shown strong psychometric properties (Langley et al., 2014).
Family Burden Assessment Scale | 5 minutes
  The Family Burden Assessment Scale (BAS) is a brief measure of subjective and objective consequences of disorder/illness on primary caretakers.
Family Accommodation Checklist and Interference Scale | 10 minutes
  The Family Accommodation Checklist and Impact Scale (FACLIS; Thompson-Hollands et al., 2014) is a parent report measure of the extent to which parents are changing their behavior in attempts to prevent or reduce child distress, and has shown strong validity and reliability in samples of youth with anxiety disorders (e.g., Thompson-Hollands et al., 2014).
Family Accommodation Scale- Anxiety | 10 minutes
  The Family Accommodation Scale-Anxiety (FASA) asks parents to rate the frequency of their participation in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety. The FASA has demonstrated strong reliability and validity (Lebowitz et al., 2013).
Working Alliance Inventory | 10 minutes
  The Working Alliance Inventory (Horvath, 1994) is a 36-item assessment of perceptions of the quality of therapeutic rapport and collaboration throughout treatment. Therapy participants and therapists will both rate each item independently on a scale from 1 (Never) to 7 (Always) to characterize their perceptions of the affective bond between the client and therapist and the extent of their agreement about the goals and tasks of treatment. The WAI has demonstrated favorable psychometric support (Horvath & Greenberg, 1989). In the present study, we will include posttreatment total scores from Mother-reports about their perceived relationship with the therapist and from Therapist-reports about their perceived relationship with the child.
Client Satisfaction Questionnaire | 3 minutes
  The Client Satisfaction Questionnaire (CSQ-8; Larsen, Attkisson, Hargreaves & Nguyen, 1979) is a generic 8-item assessment of consumer satisfaction with services received (e.g., "How would you rate the quality of the services you received?" and "If a friend were in need of similar help, would you recommend our program to him or her?"). Each item is rated on a 4-point scale and a total score is used to reflect overall satisfaction with treatment. Mother-reports at posttreatment will included in the present study. The CSQ-8 is one of the most frequently used measures of satisfaction with services and has demonstrated strong psychometric properties across a range of treatment populations.
Child Behavior Checklist | 25 minutes
  The Child Behavior Checklist (CBCL) is a standardized instrument for assessing behavioral and emotional problems, demonstrating very strong psychometric properties. Caregivers rate each item as 0 (not true), 1 (somewhat or sometimes true), or 2 (very true or often true). Empirically based scales, normed for age and gender, are generated, including three broadband dimensions (internalizing problems, externalizing problems, and total problems) as well as a number of syndrome scales and DSM-oriented scales; t-scores below 65 reflect normative functioning. For the present purposes, we will included the internalizing problems scale and the anxiety problems scale. Parents of participants ages five and below will complete the CBCL 1.5-5 (Achenbach & Rescorla, 2000) and parents of youth six and older completed the CBCL 6-18 (Achenbach, 2001).
Anxiety Disorders Interview Schedule for Children (ADIS-C/P) | 2 hours
  The ADIS is is a semi-structured diagnostic interview that assesses child psychopathology in accordance with DSM criteria.
Spence Children's Anxiety Scale | 15 minutes
  Spence Children's Anxiety Scale for Parents (SCAS-P; Spence, 1999)-a 39-item parent-report of child anxiety in youth ages 6-18-will be used to assess child anxiety in families with 6-8 year-olds. The SCAS-P has demonstrated good internal consistency, convergent validity, and discriminant validity (Nauta et al., 2004). The Total Score of the Preschool Anxiety Scale-Revised (PAS-R; Spence et al., 2008)-a 34-item parent-report of anxiety among preschoolers-will be used to assess child anxiety in families with 3-5 year-olds. The PAS-R is a downward extension of the SCAS-P for younger children and has demonstrated good construct validity and reliability (Spence et al., 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Comer, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

REFERENCES:
- [Background] Carpenter AL, Puliafico AC, Kurtz SM, Pincus DB, Comer JS. Extending parent-child interaction therapy for early childhood internalizing problems: new advances for an overlooked population. Clin Child Fam Psychol Rev. 2014 Dec;17(4):340-56. doi: 10.1007/s10567-014-0172-4. PMID 25212716
- [Background] Comer, J.S. (2015). Introduction to the special section: Applying new technologies to extend the scope and accessibility of mental health care. Cognitive and Behavioral Practice, 22, 253-257. doi:http://dx.doi.org/10.1016/j.cbpra.2015.04.002
- [Background] Comer JS, Barlow DH. The occasional case against broad dissemination and implementation: retaining a role for specialty care in the delivery of psychological treatments. Am Psychol. 2014 Jan;69(1):1-18. doi: 10.1037/a0033582. Epub 2013 Aug 5. PMID 23915401
- [Background] Comer JS, Blanco C, Hasin DS, Liu SM, Grant BF, Turner JB, Olfson M. Health-related quality of life across the anxiety disorders: results from the national epidemiologic survey on alcohol and related conditions (NESARC). J Clin Psychiatry. 2011 Jan;72(1):43-50. doi: 10.4088/JCP.09m05094blu. Epub 2010 Aug 24. PMID 20816036
- [Background] Comer JS, Furr JM, Cooper-Vince CE, Kerns CE, Chan PT, Edson AL, Khanna M, Franklin ME, Garcia AM, Freeman JB. Internet-delivered, family-based treatment for early-onset OCD: a preliminary case series. J Clin Child Adolesc Psychol. 2014;43(1):74-87. doi: 10.1080/15374416.2013.855127. Epub 2013 Dec 2. PMID 24295036
- [Background] Comer JS, Furr JM, Cooper-Vince C, Madigan RJ, Chow C, Chan P, Idrobo F, Chase RM, McNeil CB, Eyberg SM. Rationale and Considerations for the Internet-Based Delivery of Parent-Child Interaction Therapy. Cogn Behav Pract. 2015 Aug 1;22(3):302-316. doi: 10.1016/j.cbpra.2014.07.003. PMID 26120268
- [Background] Comer JS, Furr JM, Kerns CE, Miguel E, Coxe S, Elkins RM, Carpenter AL, Cornacchio D, Cooper-Vince CE, DeSerisy M, Chou T, Sanchez AL, Khanna M, Franklin ME, Garcia AM, Freeman JB. Internet-delivered, family-based treatment for early-onset OCD: A pilot randomized trial. J Consult Clin Psychol. 2017 Feb;85(2):178-186. doi: 10.1037/ccp0000155. Epub 2016 Nov 21. PMID 27869451
- [Background] Comer JS, Furr JM, Miguel EM, Cooper-Vince CE, Carpenter AL, Elkins RM, Kerns CE, Cornacchio D, Chou T, Coxe S, DeSerisy M, Sanchez AL, Golik A, Martin J, Myers KM, Chase R. Remotely delivering real-time parent training to the home: An initial randomized trial of Internet-delivered parent-child interaction therapy (I-PCIT). J Consult Clin Psychol. 2017 Sep;85(9):909-917. doi: 10.1037/ccp0000230. Epub 2017 Jun 26. PMID 28650194
- [Background] Comer JS, Puliafico AC, Aschenbrand SG, McKnight K, Robin JA, Goldfine ME, Albano AM. A pilot feasibility evaluation of the CALM Program for anxiety disorders in early childhood. J Anxiety Disord. 2012 Jan;26(1):40-9. doi: 10.1016/j.janxdis.2011.08.011. Epub 2011 Aug 25. PMID 21917417
- [Background] Costello EJ, Mustillo S, Erkanli A, Keeler G, Angold A. Prevalence and development of psychiatric disorders in childhood and adolescence. Arch Gen Psychiatry. 2003 Aug;60(8):837-44. doi: 10.1001/archpsyc.60.8.837. PMID 12912767
- [Background] Egger HL, Angold A. Common emotional and behavioral disorders in preschool children: presentation, nosology, and epidemiology. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):313-37. doi: 10.1111/j.1469-7610.2006.01618.x. PMID 16492262
- [Background] Guy, W. (1976) ECDEU Assessment Manual for Psychopharmacology - Revised. Rockville, MD: U.S. Department of Health, Education, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration, NIMH Psychopharmacology Research Branch, Division of Extramural Research Programs.
- [Background] Puliafico, A.C., Comer, J.S., & Albano, A.M. (2013). Coaching Approach behavior and Leading by Modeling: Rationale, principles, and a case illustration of the CALM Program for anxious preschoolers. Cognitive and Behavioral Practice, 20, 517-528. doi:http://dx.doi.org/10.1016/j.cbpra.2012.05.002
- [Background] Puliafico AC, Comer JS, Pincus DB. Adapting parent-child interaction therapy to treat anxiety disorders in young children. Child Adolesc Psychiatr Clin N Am. 2012 Jul;21(3):607-19. doi: 10.1016/j.chc.2012.05.005. Epub 2012 Jun 2. PMID 22800997
- [Background] Silverman, W. K., & Albano, A. M. (1997). The Anxiety Disorders Interview Schedule for children for DSM-IV: Child and parent versions. San Antonio, TX: Psychological Corporation.
- [Background] Thompson-Hollands J, Kerns CE, Pincus DB, Comer JS. Parental accommodation of child anxiety and related symptoms: range, impact, and correlates. J Anxiety Disord. 2014 Dec;28(8):765-73. doi: 10.1016/j.janxdis.2014.09.007. Epub 2014 Sep 16. PMID 25261837
- [Background] Keenan K, Wakschlag LS, Danis B. Kiddie-Disruptive Behavior Disorder Schedule. Chicago, IL: U Chicago; 2001.
- [Background] Guy W, Bonato RR. Clinical Global Impressions. Chevy Chase, MD: NIMH; 1970.
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Achenbach T, Rescorla L. Child Behavior Checklist for Ages 1.5-5. Vermont: ASEBA; 2000.
- [Background] Achenbach T. Child Behavior Checklist for Ages 6-18. Vermont: ASEBA; 2001.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Brestan E, Jacobs J, Rayfield A, Eyberg SM. (1999). A consumer satisfaction measure for parent-child treatments and its relationship to measures of child behavior change. Behav Ther. 1999;30:17-30.